CLINICAL TRIAL: NCT03187847
Title: Changes in Perceived Fatigue and Step Counts Before and After Rehabilitation. A Prospective, Single-center, Longitudinal Observational Study.
Brief Title: Rehabilitation in Multiple Sclerosis - Sometimes Too Much?
Status: Completed | Type: Observational
Sponsor: Klinik Valens (Other)
Responsible Party: Principal Investigator, Sandra Kündig, BSc in physical therapy, Klinik Valens
Other Study IDs: 2017-00728
Record Dates: First submitted 2017-05-28; First posted 2017-06-15 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Multiple Sclerosis
Keywords: Physical Activity; Fatigue; Rehabilitation
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Actigraph GT3X — The primary outcomes are measured by the Actigraph GT3X (step counts) and FSMC (fatigue scale for motor and cognitive functions questionnaire) at three different points in time (Actigraph is worn for three weeks in total).
  The secondary outcomes are emotional status, measured by the hospital anxiety and depression scale (HADS) and quality of life, measured by the Hamburg Quality of Life Questionnaire in MS (HAQUAMS).
  Other Names: FSMC; HADS

SUMMARY:
The primary objective is to evaluate changes in fatigue and physical activity (step counts) before and after rehabilitation in patients with MS (EDSS 3-6.5).

The association of changes in fatigue and physical activity will also be analyzed for disease severity (EDSS), age, emotional status (depression) of the participants.

DETAILED DESCRIPTION:
Around 2 million people worldwide have multiple sclerosis (MS) and it is the most common neurological disease in young adults. The greatest incidence of MS is found in Europe (108 per 100'000). Over 50% of the patients with MS suffer from fatigue and reduced physical activity. The association between inactivity and fatigue is low in patients with mild disability.

Rehabilitation in Valens includes intensive strength and endurance training. Endurance and walking improve in most patients, evaluated during rehabilitation with the Timed-Up and Go (TUG) and 2 minute walking tests (2MWT). However, Clinic Valens occasionally gets feedback from physical therapists in the ambulatory setting, that outcome after rehabilitation is sometimes poor and some patients with MS (pwMS) seem to be over trained, less mobile, more fatigued and need to recover for several weeks. Physical therapists in Valens know that training is fatiguing. If they knew how many, and which patients are more fatigued and less active after rehabilitation they could reduce treatment intensity and prevent overtraining.

To the knowledge of the investigators no study evaluated changes after rehabilitation in fatigue, assessed with a disease specific questionnaire (FSMC), and mobility at home using accelerometers. Potential predictors of poor outcome are disease severity (EDSS), pre-rehabilitation fatigue and depression.

The primary goal of this study therefore is to evaluate changes in fatigue and physical activity (step counts) in pwMS assessed before rehabilitation, after rehabilitation and at 2 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* EDSS 3-6.5, an EDSS 6.5 means the ability to walk 20 meters without resting, using constant bilateral assistance
* >18 years old
* German speaking
* good function of the upper extremity to put on Actigraph by themselves
* participants should be able to wear the Actigraph at least 6h/day for 7 days

Exclusion Criteria:

* inability to follow the instructions given, e.g. language problems, psychological disorders
* no informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigator plans to include at least 20 patients with multiple sclerosis with an EDSS 3-6.5, who come to Valens for rehabilitation from the end of August 2017 until July 2018.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2017-08-27 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-06-04 (Actual)

PRIMARY OUTCOMES:
Changes in Fatigue | Fatigue will be first assessed before rehabilitation in Valens, the week right after rehabilitation and at 2 months follow-up with a questionnaire given to the participant.
  The primary objective is to evaluate changes in fatigue before and after rehabilitation in patients with MS (EDSS 3-6.5). Fatigue will be assessed with the FSMC questionnaire at three different time points.
Changes in Physical Activity/Step Counts (Actigraph GT3X) | The Actigraph device will be worn for three weeks in total. Before rehabilitation (whle participants are still at home), the week right after rehabilitation and at 2 months follow up.
  The primary objective is to evaluate changes in physical activity (steps per day) before and after rehabilitation in patients with MS (EDSS 3-6.5). This will be measured by the Actigraph GT3X at three different time points.

SECONDARY OUTCOMES:
quality of life in association with changes in fatigue and physical activity | The quality of life will be assessed before rehabilitation in Valens, the week right after rehabilitation and at 2 months follow-up with a questionnaire given to the participant.
  The association of changes in fatigue and physical activity will also be analyzed for quality of life of the participants. This will be measured by the Hamburg Quality of Life Questionnaire (HAQUAMS) at three different time points.
emotional status (depression) in association with changes in fatigue and physical activity | The emotional status will be first assessed before rehabilitation in Valens, the week right after rehabilitation and at 2 months follow-up with a questionnaire given to the participant.
  The association of changes in fatigue and physical activity will also be analyzed for the emotional status of the participants. This will be measured by the hospital anxiety and depression scale (HADS) at three different time points.

OTHER OUTCOMES:
diary while wearing the Actigraph device | While measuring physical activity by the Actigraph a diary will be completed during one week before rehabilitation, the week right after rehabilitation and at 2 months follow-up
  A diary to record other activities than walking e.g. cycling, yoga, swimming will be provided during the 7 days of measurement with the Actigraph, because the device is not able to detect activities like yoga or cycling.
2 minute walking test | on the first day of rehabilitation and on the last day of rehabilitation, around 3 weeks between the two measurement time points. The rehabilitation in Valens will be planned between August 2017 and July 2018.
  2MWT (2 minute walking test) to see changes in walking speed and distance before and after rehabilitation in Valens
Timed up and Go | on the first day of rehabilitation and on the last day of rehabilitation, around 3 weeks between the two measurement time points. The rehabilitation in Valens will be planned between August 2017 and July 2018.
  TUG (timed up and go) will be assessed before and after rehabilitation to see changes in equilibrium and walking abilities

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Kündig, BSc, Principal Investigator — Klinik Valens
Locations (1):
- Kliniken Valens, Valens, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kingwell E, Marriott JJ, Jette N, Pringsheim T, Makhani N, Morrow SA, Fisk JD, Evans C, Beland SG, Kulaga S, Dykeman J, Wolfson C, Koch MW, Marrie RA. Incidence and prevalence of multiple sclerosis in Europe: a systematic review. BMC Neurol. 2013 Sep 26;13:128. doi: 10.1186/1471-2377-13-128. PMID 24070256
- [Background] Rietberg MB, van Wegen EE, Uitdehaag BM, Kwakkel G. The association between perceived fatigue and actual level of physical activity in multiple sclerosis. Mult Scler. 2011 Oct;17(10):1231-7. doi: 10.1177/1352458511407102. Epub 2011 May 17. PMID 21586484
- See also: The Atlas of MS 2013 report — https://www.msif.org/about-us/advocacy/atlas/